CLINICAL TRIAL: NCT05096546
Title: Dry Eye Cross-Sectional Study-Taiwan (DECS-TW): Observational, Multicenter, Cross-Sectional Study on Dry Eye Disease in Taiwan
Brief Title: The Proportion of Patients Diagnosed With Dry Eye by the Asia Dry Eye Society (ADES) Criteria in Taiwan (DECS-TW)
Acronym: DECS-TW
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Far Eastern Memorial Hospital (Other)
Collaborators: Santen Pharmaceutical (Taiwan) Co., LTD (Industry); Kaohsiung Medical University (Other); Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Principal Investigator, Shu-Wen Chang, Vice President, Far Eastern Memorial Hospital
Other Study IDs: FOTE-DE-01
Record Dates: First submitted 2021-10-05; First posted 2021-10-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Dry Eye Syndromes
Keywords: Dry eye disease; Asia Dry Eye Society (ADES) criteria; Taiwanese population
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group I: 1. 20 years old or older (regardless of sex)
  2. Outpatients
  3. Newly-diagnosed with dry eye disease (DED) within 6 months prior to signing the informed consent under hospital-based practice in Taiwan
  Interventions: Other: No intervention
- Group II: 1. 20 years old or older (regardless of sex)
  2. Outpatients
  3. Patients who had undergone cataract surgery and
     1. was suspected to have dry eye disease (dry eye evaluations conducted based on the routine practice) within 6 months prior to signing the informed consent or
     2. was diagnosed with dry eye disease within 6 months prior to signing the informed consent
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention will be applied for the observational study.

SUMMARY:
The study aims to determine the proportion of patients diagnosed with dry eye by the Asia Dry Eye Society (ADES) criteria, among patients diagnosed with dry eye disease under current hospital-based practice in Taiwan.

DETAILED DESCRIPTION:
This real-world, observational study aims to show in a descriptive manner to characterize the patient profile of dry eye disease in Taiwan, and to understand the local practice and its difference compared with Asia Dry Eye Society (ADES) criteria. Specific objectives include:(1) to determine the proportion of patients diagnosed with dry eye by the Asia Dry Eye Society (ADES) criteria, among patients diagnosed with dry eye disease under current hospital-based practice in Taiwan, (2) to compare the patient profile including ocular condition and dry eye-related characteristics of dry eye diagnosed with ADES criteria versus hospital-based real-world practice in Taiwan, and (3) to determine the disease characteristics of patients diagnosed with dry eye in Taiwan medical institutions.

This study will enroll patients who are diagnosed with dry eye, aged 20 years (inclusive), and are willing to provide signed informed consent. These patients will be categorized into Group I or II according to the inclusion criteria.

Clinical data of eligible patients at the time of dry eye diagnosis on medical charts will be collected. If any return visit is scheduled per routine practice before the end of data collection (Feb-28-2022), follow-up data regarding dry eye evaluations and treatments will be collected at the first follow-up visit for Group I; and within 6 months after the cataract surgery for Group II.

ELIGIBILITY:
Inclusion Criteria:

Patients who meet the criteria of either Group I OR Group II are eligible.

Group I

Patients with signed informed consent and who satisfy all of the following criteria will be included:

1. 20 years old or older (regardless of sex)
2. Outpatients
3. Newly-diagnosed with dry eye disease (DED) within 6 months prior to signing the informed consent under hospital-based practice in Taiwan

Group II

Patients with signed informed consent and who satisfy all of the following criteria will be included:

1. 20 years old or older (regardless of sex)
2. Outpatients
3. Patients who had undergone cataract surgery and

   1. was suspected to have dry eye disease (dry eye evaluations conducted based on the routine practice) within 6 months prior to signing the informed consent or
   2. was diagnosed with dry eye disease within 6 months prior to signing the informed consent

Exclusion Criteria:

Patients who meet ANY one of the following criteria are not eligible.

1. Patients who have ocular comorbidities, and appear dry eye sign and symptoms that interfere with diagnosis of dry eye disease (DED)
2. Patients who cannot confirm subjective symptoms of dry eye
3. Patients who cannot read or write, and/or could not understand dry eye questionnaire appropriately which may compromise the accuracy of questionnaire score.
4. Patients who participate in other interventional trials in the past 30 days

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: These patients will be screened in the outpatient department at Far Eastern Memorial Hospital, Kaohsiung Medical University Hospital, and Taipei Veteran General Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 540 (Estimated)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-02-28 (Actual); Study Completion 2022-07-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of patients who satisfy the criteria for dry eye disease based on the ADES criteria | At the time of dry eye diagnosis (baseline)
  The criteria are defined by Asia Dry Eye Society (ADES).

SECONDARY OUTCOMES:
Proportion of patients per dry eye severity | From baseline to 6-month follow-up
  Dry eye severity (mild, moderate, severe) is judged by the investigator.
Proportion of patients per dry eye classification | From baseline to 6-month follow-up
  Dry eye classification is judged by the investigator.
Length (mm) of soaked strip by tear for the dry eye diagnosis | From baseline to 6-month follow-up
  Unanesthetized Schirmer's test is used for assessing the tear production.
Time (second) for tear film broken with fluorescein for the dry eye diagnosis | From baseline to 6-month follow-up
  Tear break-up time (TBUT) is used to assess for tear film (evaporative dry eye disease).
Score of Ocular Surface Disease Index (OSDI) for the dry eye symptoms | From baseline to 6-month follow-up
  Ocular Surface Disease Index (OSDI) questionnaire (0 to 100 points) is used to assess the dry eye symptoms. One hundred points mean that the dry eye disease of the patient is severe.
Score of Standard Patient Evaluation of Eye Dryness (SPEED) for the dry eye symptoms | From baseline to 6-month follow-up
  Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire (0 to 28 points) is used to assess the dry eye symptoms. Twenty-eight points mean that the symptoms of dry eye disease is severe.
Visual analogue scale (VAS) for the dry eye severity | From baseline to 6-month follow-up
  Visual analogue scale (VAS) (0 to 10 [mild to severe]) is used to assess the dry eye severity based on the symptoms.
Difference in length (mm) of soaked strip by tear between patients who satisfy the criteria for dry eye disease based on the ADES consensus report and the whole population (i.e., hospital-based real-world practice) | At the time of dry eye diagnosis (baseline)
  Unanesthetized Schirmer's test is used for assessing the tear production.
Difference in time (second) for tear film broken with fluorescein between patients who satisfy the criteria for dry eye disease based on the ADES consensus report and the whole population (i.e., hospital-based real-world practice) | At the time of dry eye diagnosis (baseline)
  Tear break-up time (TBUT) is used to assess for tear film (evaporative dry eye disease).
Difference in score of Ocular Surface Disease Index (OSDI) between patients who satisfy the criteria for dry eye disease based on the ADES consensus report and the whole population (i.e., hospital-based real-world practice) | At the time of dry eye diagnosis (baseline)
  Ocular Surface Disease Index (OSDI) questionnaire (0 to 100 points) is used to assess the dry eye symptoms. One hundred points mean that the dry eye disease of the patient is severe.
Difference in score of Standard Patient Evaluation of Eye Dryness (SPEED) between patients who satisfy the criteria for dry eye disease based on the ADES consensus report and the whole population (i.e., hospital-based real-world practice) | At the time of dry eye diagnosis (baseline)
  Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire (0 to 28 points) is used to assess the dry eye symptoms. Twenty-eight points mean that the symptoms of dry eye disease is severe.
Difference in visual analogue scale (VAS) between patients who satisfy the criteria for dry eye disease based on the ADES consensus report and the whole population (i.e., hospital-based real-world practice) | At the time of dry eye diagnosis (baseline)
  Visual analogue scale (VAS) (0 to 10 [mild to severe]) is used to assess the dry eye severity based on symptoms.
Proportion of patients who do not satisfy the criteria for dry eye disease based on the ADES per dry eye severity | From baseline to 6-month follow-up
  Dry eye severity (mild, moderate, severe) is judged by the investigator.
Proportion of patients who do not satisfy the criteria for dry eye disease based on the ADES per dry eye classification | From baseline to 6-month follow-up
  Dry eye classification is judged by the investigator.
Length (mm) of soaked strip by tear using unanesthetized Schirmer test of patients who do not satisfy the criteria for dry eye disease based on the ADES | From baseline to 6-month follow-up
  Schirmer's test is used for assessing the tear production.
Time (second) for tear film broken with fluorescein of patients who do not satisfy the criteria for dry eye disease based on the ADES | From baseline to 6-month follow-up
  Tear break-up time (TBUT) is used to assess for tear film (evaporative dry eye disease).
Score of Ocular Surface Disease Index (OSDI) of patients who do not satisfy the criteria for dry eye disease based on the ADES | From baseline to 6-month follow-up
  Ocular Surface Disease Index (OSDI) questionnaire (0 to 100 points) is used to assess the dry eye symptoms. One hundred points mean that the dry eye disease of the patient is severe.
Score of Standard Patient Evaluation of Eye Dryness (SPEED) of patients who do not satisfy the criteria for dry eye disease based on the ADES | From baseline to 6-month follow-up
  Standard Patient Evaluation of Eye Dryness (SPEED) questionnaire (0 to 28 points) is used to assess the dry eye symptoms. Twenty-eight points mean that the symptoms of dry eye disease is severe.
Visual analogue scale (VAS) of patients who do not satisfy the criteria for dry eye disease based on the ADES | From baseline to 6-month follow-up
  Visual analogue scale (VAS) (0 to 10 [mild to severe]) is used to assess the dry eye severity based on the symptoms.

CONTACTS AND LOCATIONS:
Locations (3):
- Taiwan (3):
  - Kaohsiung Medical University Hospital, Kaohsiung City
  - Far Eastern Memorial Hospital, New Taipei City
  - Taipei Veteran General Hospital, Taipei

IPD SHARING:
Plan to Share IPD: No